CLINICAL TRIAL: NCT01055964
Title: a Comparative Pharmacokinetic Study of Two Oral Formulations of Tacrolimus in Renal Allograft Recipients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jongwon Ha, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: Tacrobell-01
Record Dates: First submitted 2010-01-24; First posted 2010-01-26 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Pharmacokinetics; Tacrolimus
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tacrobell (Experimental)
  Interventions: Drug: Tacrolimus
- Prograf (Active Comparator)
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus

SUMMARY:
The aim of this study is to identify the pharmacokinetic differences between two oral forms of Tacrolimus and consequent nephrotoxicity.

ELIGIBILITY:
Inclusion Criteria:

* ABO-compatible renal transplant recipients

Exclusion Criteria:

* multi-organ transplant
* HIV(+) donor or recipients
* history of malignancy other than skin cancer (except completely cured basal cell ca or squamous cell ca)
* more than three-fold increase in AST or ALT level for 28 days
* pregnancy
* lactation

Ages: 19 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2008-09; Primary Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
pharmacokinetics | at postoperative 10~14 days and at postoperative 6 months for crossover study

CONTACTS AND LOCATIONS:
Overall Officials: Jongwon Ha, MD, PhD, Principal Investigator — Seoul National University
Locations (1):
- Seoul National University Hospital, Seoul, South Korea